CLINICAL TRIAL: NCT06695390
Title: Development of Humanistic Care Competencies Scale for Nursing Students
Brief Title: Scale Development Study
Status: Completed | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Aysun Acun 8
Record Dates: First submitted 2024-10-24; First posted 2024-11-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-10

CONDITIONS: Nursing Students
Keywords: humanistic care; Nursing students; care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Nursing students' humanistic care competence — A cross-sectional study with nursing students

SUMMARY:
The aim of this study was to develop a scale to measure humanistic care competencies for nursing students.

DETAILED DESCRIPTION:
Studies in the literature show that humanistic care perception should develop as a student. At this point, it is of great importance to know the competency level of nursing students regarding humanistic care. Although the evaluation of competency and professional development is an important point in nursing education, the difficulty of defining the concept of competency reveals the need for measurement tools. A valid and reliable scale is needed to be used in measuring the humanistic care competencies of nursing students. Reliable measurement of humanistic care competency in nursing students will guide the education curriculum. This study is an original study in its field as it is the development of a scale measuring competency regarding humanistic care.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate.
* Being a 2nd, 3rd or 4th grade student in the nursing department.

Exclusion Criteria:

* Being a first year student.
* Being absent and on academic leave during the period in which the study was conducted.

Ages: 17 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 340 stduents
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Information questionnaire on socio-demographic characteristics of nursing students | 12/11/2024-20/11/2024
  Descriptive information
Scale questionnaire measuring humanistic care competence of nursing students | 01/11/2024-01/12/2024
  Nursing students and care

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)